CLINICAL TRIAL: NCT05829460
Title: Primary Prevention and Uterine Preservation in Premenopausal Women With Obesity and Endometrial Hyperplasia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202402083
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — semaglutide; Progestins

STUDY DESIGN:
Intervention Model Description: Patients will be randomized on a 1:1 basis to either progestin + semaglutide 2.4 mg or progestin + placebo. Randomization will be stratified by previous progestin and metformin use.
Who Masked: Participant, Care Provider
Masking Description: Participant and pathologist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Semaglutide + progestin (Experimental): * The progestin will be delivered via the levonorgestrel-releasing IUD and it is standard of care.
  * Will receive injectable pens containing semaglutide and will be self-administered on a weekly basis for up to 104 weeks. Dosing will be escalated during weeks 1 through 16 (start at 0.25 mg up to 2.4 mg).
  * Will be enrolled in a behavioral weight program that is optional to attend. The program will be delivered in a closed-group format. The group program will consist of 12 consecutive 60 minute weekly visits, and will recur every three months such that participants can join the soonest available Week 1 session after study enrollment. Each group session will focus on providing education and cognitive/behavioral strategies to achieve a healthier, reduced-calorie diet and a more physically active lifestyle. Cognitive/behavioral strategies will consist of goal setting, problem solving, cognitive restructuring, stimulus control, and stress management.
  Interventions: Drug: Semaglutide; Drug: LNG-IUD (Progestin); Behavioral: Telemedicine behavioral weight program
- Arm 2: Placebo + Progestin (Active Comparator): * The progestin will be delivered via the levonorgestrel-releasing IUD and it is standard of care.
  * Will receive injectable pens containing the placebo and will be self-administered on a weekly basis for up to 104 weeks.
  * Will be enrolled in a behavioral weight program that is optional to attend. The program will be delivered in a closed-group format. The group program will consist of 12 consecutive 60 minute weekly visits, and will recur every three months such that participants can join the soonest available Week 1 session after study enrollment. Each group session will focus on providing education and cognitive/behavioral strategies to achieve a healthier, reduced-calorie diet and a more physically active lifestyle. Cognitive/behavioral strategies will consist of goal setting, problem solving, cognitive restructuring, stimulus control, and stress management.
  Interventions: Drug: Placebo; Drug: LNG-IUD (Progestin); Behavioral: Telemedicine behavioral weight program

INTERVENTIONS:
Drug: Semaglutide — This medication is self-administered as a subcutaneous injection in the abdomen, thigh, or upper arm; injection site should be rotated when using the same body region.
  Arms: Arm 1: Semaglutide + progestin
Drug: Placebo — This medication is self-administered as a subcutaneous injection in the abdomen, thigh, or upper arm; injection site should be rotated when using the same body region.
  Arms: Arm 2: Placebo + Progestin
Drug: LNG-IUD (Progestin) — Released via the levonorgestrel-releasing IUD.
Behavioral: Telemedicine behavioral weight program — Optional to attend.

SUMMARY:
The investigators hypothesize that combined treatment with the GLP-1R agonist semaglutide 2.4 mg and levonorgestrel intrauterine device (LNG-IUD), compared to LNG-IUD alone, will result in improved likelihood of uterine preservation, sustained weight loss, improved endometrial and metabolomic response to progestin, and improved quality of life in premenopausal women with endometrial hyperplasia who desire uterine preservation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed non-atypical endometrial hyperplasia (EH) or complex atypical endometrial hyperplasia (AEH).

  * Patients with a previous diagnosis of EH or AEH who are already being followed with conservative management with oral or LNG-IUD progestin therapy are eligible provided they have not previously been on a GLP-1R agonist within 3 months prior to enrollment.
  * For patients with a previous diagnosis of EH or AEH who have been placed on progestin prior to study entry, the duration of IUD or oral progestin use prior to trial entry should be less than or equal to 6 months.
* Premenopausal woman with a uterus.
* At least 18 years of age and no more than 45 years of age.
* Interested in uterine preservation/fertility-sparing treatment.
* BMI ≥ 30 kg/m2.
* Prior or current receipt of progestin is allowed as above. Willingness to undergo placement of LNG-IUD at the time of study entry.
* Prior or current receipt of metformin is allowed.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Prior use of GLP-1 receptor agonist (exenatide, liraglutide, or other) or pramlintide or any DPP-4 inhibitor in the 3 months prior to date of registration.
* History of type 1 diabetes.
* History of type 2 diabetes requiring use of insulin.
* Acute decompensation of glycemic control.
* Concomitant use of other weight management drugs or drugs for short-term weight loss.
* History of surgery or use of a device to treat obesity.
* Uncontrolled thyroid disease
* Acute coronary or cerebrovascular event in the previous 60 days.
* Currently planned coronary, carotid, or peripheral artery revascularization.
* Chronic heart failure (NYHA class IV).
* Evidence of renal dysfunction as defined by creatinine clearance < 60 ml/minute.
* History of solid organ transplant or awaiting solid organ transplant.
* Diagnosis of any malignant neoplasm or current, active treatment with chemotherapy or radiation.
* Family or personal history of multiple endocrine neoplasia syndrome type 2 (MEN 2) or familial medullary thyroid carcinoma (MTC).
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to progestin, semaglutide, or other agents used in the study.
* History of diabetic retinopathy.
* Recent history of pancreatitis, defined as less than 6 months prior to enrollment.
* History of suicidal attempts or active suicidal ideation.
* Significant active psychiatric disease, including recent psychiatric inpatient admission or use of any psychiatric medications that are not stabilized.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Participants must have a negative serum pregnancy test within 7 days of date of registration.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL, they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration, or they are receiving anti-retrovirals that affect progestin levels. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with endometrial hyperplasia free biopsy with uterine preservation | At 2 years (or exit from study)

SECONDARY OUTCOMES:
Time to resolution of endometrial hyperplasia (EH) | Through completion of follow-up (estimated to be 4 years)
Change in weight | From baseline to 2 years
Change in Cancer Worry Impact of Events Scale (CWIES) | At enrollment, 12 months, and end of treatment (estimated to be 2 years)
  The CWIES is a 15-item self-report measure evaluating stress reactions and traumatic experiences, specifically inquiring about cancer worry-specific distress. Range of values for each individual item will be a Likert Scale from 0-5. 0=not at all and 5=often. The higher the score, the more cancer-worry specific distress the participant has.
Change in Impact of Weight on Quality of Life (IWQOL-Lite) | At enrollment, 12 months, and end of treatment (estimated to be 2 years)
  The IWQOL-Lite provides a total score and scores for five subscales: physical function, self-esteem, sexual life, public distress and work. Scores range from 0 to 100 with lower scores indicating greater impairment.
Hyperplasia-free survival | Through completion of follow-up (estimated to be 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea R Hagemann, M.D., MSCI, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu